CLINICAL TRIAL: NCT06107127
Title: 2 RCTS: Investigate the Relationship Between Pain-free Shoulder Abduction and External Rotation Force and Pain and Disability - Assess the Effectiveness of Two Different Forms of Exercise Treatment
Brief Title: STOP - START With Rotator Cuff-related Shoulder Pain (RCRSP) Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sussex Community NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 331819
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Musculoskeletal Diseases
Keywords: rotator cuff
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Researcher 1 (Active Comparator): Using their symptomatic arm participants will be asked to push against a fixed force dynamometer (hand held force gauge), starting with a low level of effort and gradually increasing their effort stopping either at the point that they start to feel pain or when they feel they have pushed as forcefully as they can.
  Interventions: Procedure: STOP
- Researcher 2 (Active Comparator): Using their symptomatic arm participants will be asked to push against a fixed force dynamometer (hand held force gauge), starting with a low level of effort and gradually increasing their effort stopping either at the point that they start to feel pain or when they feel they have pushed as forcefully as they can.
  Interventions: Procedure: STOP

INTERVENTIONS:
Procedure: STOP — Using their symptomatic arm participants will be asked to push against a fixed force dynamometer (hand held force gauge), starting with a low level of effort and gradually increasing their effort stopping either at the point that they start to feel pain or when they feel they have pushed as forcefully as they can.

SUMMARY:
Shoulder pain is the third most common type of musculoskeletal (MSK) disorder for which people seek medical care. Roughly 70% of all shoulder pain can be accounted for by one condition, namely rotator ruff-related shoulder pain (RCRSP). Despite limited research it is thought that a lack of pain-free force production of certain shoulder muscles is a key finding in those with RCRSP. Strengthening exercise appears to be an important treatment for RCRSP. However, there remains uncertainty regarding the optimal choice of exercise. It has been suggested essential to target the rotator cuff muscles. Despite this claim, exercise specific to these muscles has not been compared to exercise that specifically avoids significant rotator cuff recruitment. A clearer understanding could result in more effective treatment, and improved exercise adherence.

Key questions that this research aims to answer are:

1. Is it important to measure pain-free force when treating people with RCRSP?
2. Is it more effective to target the rotator cuff muscles than not when using exercise to treat RCRSP? To attempt to answer these questions this study will be split into two trials. Patients referred to Sussex Community NHS Foundation trust for treatment of RCRSP will be screened by a Physiotherapist for eligibility and those interested will be asked to give consent to participate. Trial 1 will involve participants attending a one-off 45-minute assessment. Data collection will run over a 6-month period. Participants in Trial 2 will be required to attend a minimum of 10 (or maximum of 12) 45-minute exercise sessions over a 12-16-week period. Trail 2 will last approximately 18 months, with outcomes being recorded when participants finish their exercise sessions and at 6 and 12 months after the date they started the trial.

DETAILED DESCRIPTION:
The aims of this study are to

1. investigate the relationship between pain-free shoulder abduction and external rotation force and pain and disability in those with RCRSP, and
2. to assess the effectiveness of two different forms of exercise aimed at reducing pain and disability in patients with RCRSP.

The key questions that this research aims to answer are:

1. Is pain-free shoulder force testing in patients with RCRSP using portable hand-held dynamometer reliable?
2. Do reductions in pain-free force using this method correlate with severity of shoulder pain and disability?
3. When treating RCRSP using resistance training (RT) exercise to specifically target the rotator cuff is compared to resistance training designed to avoid a significant contribution from these muscles, are there differences in outcome?
4. What factors might mediate the changes in outcome in these two groups? The design is a randomised controlled trial. Trial 1 Participants will be allocated to one of two groups. Group one will be allocated researcher no. one and group two will be allocated to researcher no. two. Relevant tests will then be carried out. The two groups will then swap researcher and be tested again. The test: Using their symptomatic arm participants will be asked to push against a fixed force dynamometer (hand held force gauge), starting with a low level of effort and gradually increasing their effort stopping either at the point that they start to feel pain or when they feel they have pushed as forcefully as they can. Participants will be advised to rest for 1 minute before repeating this process a total of three times. All three measures will be recorded, and a mean will be calculated. The same procedure will then be carried out on their asymptomatic shoulders. A ten-minute break will follow, and the process will be repeated with the second assessor. This ensures that the order in which patients are assessed cannot influence the results. Once measured, the difference in pain-free force between symptomatic and asymptomatic shoulders will be described in terms of an index (a score reported as a percentage). Outcome measures will be taken once the session is over. Pain-free shoulder force index. Shoulder pain and disability index. Trial 2 Participants will be allocated in to one of the two exercise programme intervention groups. Participants will be asked to complete a minimum of ten sessions of exercise over a sixteen week period from when they start.

Group 1 - Participants will perform resistance exercises that involve pushing against a weighted pulley machine.

Exercise intensity will be progressed over each session as participants become accustomed to the stimulus involved.

Group 2 - Participants will perform resistance exercises that involve pulling against a weighted pulley machine.

Exercise intensity will be progressed over each session as participants become accustomed to the stimulus involved. Outcome measures will be taken once all sessions have been completed, and at 6 and 12 months.

Outcome measures are: Shoulder pain and disability index. Pain-free shoulder force index (if considered reliable during Trial 1).

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 years or older

  * Shoulder pain of at least 3-month duration.
  * Minimal resting pain
  * Pain reproduced during resisted testing in shoulder abduction and/or external rotation.
  * Diagnosis of rotator cuff-related shoulder pain (RCRSP) suggested by at least 3 of the following tests being positive:

    1. Near normal passive range of shoulder flexion / abduction / external rotation
    2. Pain may or may not be present during active shoulder external rotation when tested at 0° of shoulder abduction but will increase with resisted* external rotation.
    3. Pain may or may not be present during active shoulder external rotation when tested at 90° of shoulder abduction but will increase with resisted external rotation.
    4. Pain may or may not be present during active shoulder abduction when tested through range but will increase with resisted abduction (plane of scapula, elbow extended, forearm in mid prone) at 45° and / or 90° and / or 150° and / or end-range.
    5. Pain may or may not be present during active shoulder flexion when tested through range but will increase with resisted flexion (elbow extended, forearm in mid prone) at 45° and / or 90° and / or 150° and / or end-range.
    6. Presence of a painful arc of movement.

Exclusion Criteria:

* Known calcific tendinopathy, based on previous imaging.

  * Patients with clinical signs of massive rotator cuff tears as defined by presence of gross weakness of rotator cuff muscles in the absence of pain.
  * Other shoulder disorders e.g., frozen shoulder, severe osteoarthritis, fracture, acromioclavicular joint pathology, history of shoulder dislocation.
  * Shoulder external rotation less than 45 degrees or 50% of the opposite side.
  * Undergone previous shoulder surgery on same side.
  * Symptomatic cervical spine pathology, defined as reproduction of neck, shoulder or upper limb symptoms with active physiological cervical spine movement of any of the following movements in isolation or in combination: flexion, extensions: rotation (left and / or right), side flexion (left and / or right).
  * Presence of significant co-morbidity e.g., neurological disorders, rheumatoid arthritis, unstable diabetes, unstable blood pressure
  * Current carcinoma, TB, or HIV
  * Unlikely to be able to perform required clinical assessment tasks.
  * Inability to understand written or spoken English language.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index | 10 to 12 weeks
  The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability.